CLINICAL TRIAL: NCT06282770
Title: Utilizing Photobiomodulation Via Laser Diode Belts To Treat Chronic Lower Back Pain in Patients Who Have Undergone Spinal Fusion and Decompression Surgery
Brief Title: Photobiomodulation for Lower Back Pain Post Spinal Fusion and Decompression Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel Lu, MD, PhD, Neurosurgeon, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB#23-000444
Record Dates: First submitted 2023-05-23; First posted 2024-02-28 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Spinal Fusion; Chronic Lower Back Pain
Keywords: Photobiomodulation; Laser Diode; Inflammation; Spinal Fusion; Spinal Decompression; Lumbar; Back Pain
MeSH Terms: conditions — Inflammation; Back Pain

STUDY DESIGN:
Intervention Model Description: Participants are assigned in parallel to one of two arms (active photobiomodulation brace or sham brace). Assignment occurs once prior to surgery and remains fixed for the duration of the 12-week study. There is no crossover between arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants in this study will not be told which belt is the sham diode brace or which is the functional diode brace. The assessor of the study will also be blinded to which belt each subject has, and data will be analyzed blindly based on patient ID alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Brace With Electrical Diodes (Experimental): The patient will be given a laser diode brace to wear for 1 year. At the defined time points following surgery (2, 4, 6, 8, and 12 weeks), subjects will be asked to complete pain and ability-to-function questionnaires and submit scar/wound images to determine their status at each time interval.
  Interventions: Device: Laser Diode Brace
- Sham Brace Without Electrical Diodes (Sham Comparator): The patient will be given a sham/placebo laser diode brace to wear for 1 year. At the defined time points following surgery (2, 4, 6, 8, and 12 weeks), subjects will be asked to complete pain and ability-to-function questionnaires and submit scar/wound images to determine their status at each time interval.
  Interventions: Device: Sham Laser Diode Brace

INTERVENTIONS:
Device: Laser Diode Brace — The device is a brace with laser diodes. The braces light up and the red light has therapeutic abilities.
  Other Names: Laser Brace
  Arms: Brace With Electrical Diodes
Device: Sham Laser Diode Brace — The Sham brace has no therapeutic ability and will act as a placebo.
  Other Names: Shame Brace
  Arms: Sham Brace Without Electrical Diodes

SUMMARY:
After spinal fusion and decompression surgery there is a possible risk of developing chronic back pain. After surgery there is typically inflammation around the operation site and this inflammation can be painful and debilitating to patients.

Many possible treatment plans have been incorporated to assist the patient with recovery - notably medications, physical therapy, and braces. However, few studies have looked at laser diodes that utilize high-power laser lights that are aimed at decreasing pain and inflammation. Investigators aim to look compare patients using a back brace with laser diodes within versus those who wear a normal brace used as a placebo. Investigators will also assess the patient's surgical wound to monitor the progression of wound healing while using the brace.

DETAILED DESCRIPTION:
This study will review charts of 80 patients who have experienced chronic back pain at various operative sites of a teaching medical institution, including the inpatient academic medical center, outpatient ambulatory hospital, and regional trauma center. Deidentified demographic data that will be collected via extensive chart reviews include age, sex, BMI, preoperative diagnosis, pre- and post-operative pain scales, motor exams, and function questionnaires. Operative data will include operative time and estimated blood loss (EBL).

Patients that have already expressed interest in receiving spinal fusion or decompression surgery will come into clinic for consultation and enrollment in the study. Regardless of study participation, patients will receive either surgery. For the study, 80 subjects will be enrolled (40 with minimally invasive spinal fusion and 40 with minimally invasive decompression surgeries). Prior to the surgery date, subjects will complete pre-operation questionnaires that include the Visual Analogue Scale (VAS) and the Oswestry-Low-Back-Pain-Disability Index (ODI) to self-evaluate their current pain level and ability to perform basic lifestyle functions, respectively. Following surgery, enrolled subjects will then receive a brace that contains laser diodes or a sham (placebo) brace that appears identical to the diode-containing brace but lacks functional diodes. Subjects will wear the brace 3 times/day for 12 minutes each session for 12 weeks. They will complete and submit via the REDCap electronic submission portal the VAS and ODI questionnaires at the following time points after surgery: 2, 4, 6, 8, and 12 weeks. Subjects will also submit photos of their surgical scars for evaluation by the research study team members. Scar and wound healing will be assessed using image analysis software (Image J) according to the Stony Brook Scar Evaluation scale. Photos will be stored on a safe and secure encrypted server.

ELIGIBILITY:
Inclusion Criteria:

* Subject will have undergone minimally invasive spinal fusion surgery or spinal decompression surgery in their lower back L1-S1.
* Have low back pain of >3 months and a pain threshold of > 4 (as described by the the subject), age > 18 years, and English speaking to eliminate possible miscommunication and consequent human error regarding belt use.
* Subject must have had surgery at minimum to 1 year prior to start of study and no more than 5 years prior to start to study

Exclusion Criteria:

* Patients with tumors
* Current infection
* Drug misuse history
* Skin conditions preclude the use of laser belt
* Severe spondylolisthesis, spondylolysis, spinal stenosis, ankylosing spondylitis
* Previous low back surgery exceeding 5 years to initial start date.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported patient outcome questionnaires after photobiomodulation therapy - VAS | 3 months
  Subjects will fill out two questionnaires related to their pain and quality of life before and after surgery with laser diode brace photobiomodulation therapy.
  The first survey is the Visual Analog Scale (VAS), which asks subjects to state how good or bad their current health state is on a scale of 0-100, 1 being the worst imaginable health state and 100 being the best imaginable health state. There are two additional questions that ask subjects to provide a rate their current back and leg pain on a scale of 0-10, with 0 being no pain and 10 being worst imaginable pain.
Self-reported patient outcome questionnaires after photobiomodulation therapy - ODI | 3 months
  The second survey is the Oswestry Disability Index (ODI), which is designed to provide information on how the subject's pain is affecting their everyday life. There are 10 sections on the survey each graded on a scale from 0-5 with 5 being the most impaired. The total score scales from 0-50, where 0-10 denotes minimal disability and 40-50 denotes that the pain impinges on all aspects of their daily lives.

SECONDARY OUTCOMES:
Stony Brook Scar Evaluation | 3 months
  Surgical scar healing will be examined to see if there is any promotion of wound healing due to the therapeutic advantage from the brace photobiomodulation therapy. Assessments include scar/wound size (in mm) and scar/wound healing using the Image J software.
  The Stony Brook Scar Evaluation will score the scar from 0-5 where 5 shows significant healing.

CONTACTS AND LOCATIONS:
Overall Officials: Sara K Chung, PA, Study Director — University of California, Los Angeles; Sandra M Holley, PhD, Study Director — University of California, Los Angeles; Sichen Li, PhD, Study Director — University of California, Los Angeles; Adreanne Rivera, BS, Study Director — University of California, Los Angeles
Locations (2):
- United States (2):
  - Semel Institute of Neuroscience at UCLA, Los Angeles, California
  - UCLA Clinical and Translational Research Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No